CLINICAL TRIAL: NCT00995904
Title: A Randomized, Open-Label, 3-Dose, 3-Period, Crossover Phase 2 Study Investigating the Tolerability and Pharmacokinetics of MAP0010 in Children 4 Through 11 Years Old With a History of Mild-To-Moderate Stable Asthma
Brief Title: Tolerability and PK of Submicron Budesonide in Children 4 to 11 Years Old With Mild-To-Moderate Stable Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAP0020-CL-P201
Record Dates: First submitted 2009-10-06; First posted 2009-10-15 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: asthmatic children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A, then Treatment B, then Treatment C (Experimental): Study visits were separated by 3-7 day intervals. Treatment A: 84ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 4
  Interventions: Drug: 84ug MAP0020; Drug: 42ug MAP0020; Drug: 21ug MAP0020
- Treatment A, then Treatment C, then Treatment B (Experimental): Study visits were separated by 3-7 day intervals. Treatment A: 84ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 4
  Interventions: Drug: 84ug MAP0020; Drug: 42ug MAP0020; Drug: 21ug MAP0020
- Treatment B, then Treatment A, then Treatment C (Experimental): Study visits were separated by 3-7 day intervals. Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment A: 84ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 4
  Interventions: Drug: 84ug MAP0020; Drug: 42ug MAP0020; Drug: 21ug MAP0020
- Treatment B, then Treatment C, then Treatment A (Experimental): Study visits were separated by 3-7 day intervals. Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment A: 84ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) at Visit 4
  Interventions: Drug: 84ug MAP0020; Drug: 42ug MAP0020; Drug: 21ug MAP0020
- Treatment C, then Treatment A, then Treatment B (Experimental): Study visits were separated by 3-7 day intervals.
  Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment A: 84ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 4
  Interventions: Drug: 84ug MAP0020; Drug: 42ug MAP0020; Drug: 21ug MAP0020
- Treatment C, then Treatment B, then Treatment A (Experimental): Study visits were separated by 3-7 day intervals. Treatment C: 21ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) at Visit 2; Treatment B: 42ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) at Visit 3; Treatment A: 84ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) at Visit 4
  Interventions: Drug: 84ug MAP0020; Drug: 42ug MAP0020; Drug: 21ug MAP0020

INTERVENTIONS:
Drug: 84ug MAP0020 — 84ug of unit dose budesonide inhalation suspension delivered by Aeroneb® Go (MAP0020) as per protocol
Drug: 42ug MAP0020 — 42ug of unit dose budesonide inhalation suspension delivered by Aeroneb® Go (MAP0020) as per protocol
Drug: 21ug MAP0020 — 21ug of unit dose budesonide inhalation suspension delivered by Aeroneb® Go (MAP0020) as per protocol

SUMMARY:
This Phase 2 study was to investigate the tolerability of unit dose budesonide (MAP0020) at three doses in pediatric volunteers with a diagnosis and history of mild-to-moderate stable asthma and evaluate the pharmacokinetic profile of budesonide resulting from inhalation aerosol delivery.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female children with a documented diagnosis of mild-to-moderate persistent asthma (according to the 2007 NIH [EPR] criteria) for at least 1 year prior to screening and medically stable for a minimum of 6 months prior to screening.
2. Children 4 through 11 years old (up to one day prior to their 12th birthday at randomization).
3. Body weight >=45 lbs, body mass index (BMI) <=30 kg/m2
4. ICS users had to have been taking an ICS for >=3 months and on a stable dose for >= 1 month before Visit 1.ICS users had to be stable enough and able to withhold their therapeutic ICS for 24 hours prior to study drug administration,
5. Subjects already on stable immunotherapy (ie, allergy shots)if not anticipated to change during the study.

Key Exclusion Criteria:

1. Females of child-bearing potential/menarche.
2. Diagnosis of any other significant chronic illness or abnormality.
3. Use of corticosteroids

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ratner, MD, Principal Investigator — Sylvana Research Associates; Ammar Hatab, MD, Principal Investigator — West Coast Clinical Trials LLC
Locations (2):
- United States (2):
  - West Coast Clinical Trials LLC, Cypress, California
  - Sylvana Research Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 3-treatment, 3-period, 6-sequence crossover study. Each subject received all 3 treatments in a randomly assigned order: treatments A, B, and C, the sequences were ABC, ACB, BAC, BCA, CAB, and CBA.
Groups:
- Treatment B, Then Treatment C, Then Treatment A: Study visits were separated by 3-7 day intervals. Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment A: 84ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 4
- Treatment C, Then Treatment B, Then Treatment A: Study visits were separated by 3-7 day intervals. Treatment C: 21ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 2; Treatment B: 42ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 3; Treatment A: 84ug MAP0020 (unit dose budesonide delivered by Aeroneb® Go) at Visit 4
Period: Visit 2 (Randomization)
Arm/Group | Treatment A, Then Treatment B, Then Treatment C | Treatment A, Then Treatment C, Then Treatment B | Treatment B, Then Treatment A, Then Treatment C | Treatment B, Then Treatment C, Then Treatment A | Treatment C, Then Treatment A, Then Treatment B | Treatment C, Then Treatment B, Then Treatment A
Started | 4 | 3 | 4 | 5 | 5 | 4
Completed | 4 | 3 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 3
Arm/Group | Treatment A, Then Treatment B, Then Treatment C | Treatment A, Then Treatment C, Then Treatment B | Treatment B, Then Treatment A, Then Treatment C | Treatment B, Then Treatment C, Then Treatment A | Treatment C, Then Treatment A, Then Treatment B | Treatment C, Then Treatment B, Then Treatment A
Started | 4 | 3 | 4 | 5 | 5 | 3 (One subject was withdrawn from the study after completion of Visit 2 but prior to Visit 3.)
Completed | 4 | 3 | 4 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 4
Arm/Group | Treatment A, Then Treatment B, Then Treatment C | Treatment A, Then Treatment C, Then Treatment B | Treatment B, Then Treatment A, Then Treatment C | Treatment B, Then Treatment C, Then Treatment A | Treatment C, Then Treatment A, Then Treatment B | Treatment C, Then Treatment B, Then Treatment A
Started | 4 | 3 | 4 | 5 | 5 | 3
Completed | 4 | 3 | 4 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Visit (Final Visit)
Arm/Group | Treatment A, Then Treatment B, Then Treatment C | Treatment A, Then Treatment C, Then Treatment B | Treatment B, Then Treatment A, Then Treatment C | Treatment B, Then Treatment C, Then Treatment A | Treatment C, Then Treatment A, Then Treatment B | Treatment C, Then Treatment B, Then Treatment A
Started | 4 | 3 | 4 | 5 | 5 | 3
Completed | 4 | 3 | 4 | 5 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients that were enrolled in the study.
Arm/Group | All Patients
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (1.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Budesonide After Administration of MAP0020
Description: The maximum concentration (Cmax) is the highest concentration of a drug measured in the plasma. Plasma is the clear portion of the blood. The Cmax of Budesonide is reported in picograms per milliliter (pg/ml).
Time Frame: 12 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- 21ug MAP0020: 21ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) as per protocol
- 42ug MAP0020: 42ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) as per protocol
- 84ug MAP0020: 84ug of unit dose budesonide delivered by Aeroneb® Go (MAP0020) as per protocol
Arm/Group | 21ug MAP0020 | 42ug MAP0020 | 84ug MAP0020
Number analyzed (Participants) | 22 | 22 | 22
pg/ml | 92.5 (72.9) | 175 (96.0) | 370 (236)

2. Primary Outcome: AUC(0-inf) of Budesonide After Administration of MAP0020
Description: The AUC(0-inf) is the area under the plot of plasma concentration of drug to time infinity after drug administration. Budesonide AUC(0-inf) is reported in picograms times minutes per milliliter (pg*min/ml).
Time Frame: 12 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: pg*min/ml
Arm/Group | 21ug MAP0020 | 42ug MAP0020 | 84ug MAP0020
Number analyzed (Participants) | 22 | 22 | 22
pg*min/ml | 3750 (1560) | 8710 (3270) | 19400 (8230)

3. Primary Outcome: Half-life (t1/2) of Budesonide After Administration of MAP0020
Description: Half-life (t1/2) is the time for the drug to decrease to half of its maximum concentration. Budesonide t1/2 is reported in minutes.
Time Frame: 12 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 21ug MAP0020 | 42ug MAP0020 | 84ug MAP0020
Number analyzed (Participants) | 22 | 22 | 22
minutes | 53.3 (31.2) | 74.6 (29.8) | 86.9 (29.0)

ADVERSE EVENTS:
Description: All 25 subjects who received 21ug MAP0020, 24 subjects who received 42ug MAP0020, and 24 subjects who received 84ug MAP0020 are included in the adverse event analysis.
Arm/Group | 21ug MAP0020 | 42ug MAP0020 | 84ug MAP0020
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/25 | 1/24 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 21ug MAP0020 (N=25) | 42ug MAP0020 (N=24) | 84ug MAP0020 (N=24)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.